CLINICAL TRIAL: NCT03864588
Title: A Randomized Controlled Trial Comparing Intraoperative Surgeon-Performed Versus Anesthesiologist-Performed Adductor Canal Blockade After Primary Total Knee Arthroplasty
Brief Title: Comparing Ropivacaine Adductor Canal Blockade by Surgeon Versus Anesthesiologist
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: Sharpe-Strumia Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018LonnerSS
Record Dates: First submitted 2018-10-26; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Pain, Postoperative; Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Personal Satisfaction | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Anesthesiologist preforms ultrasound guided adductor canal block post-operatively
  Interventions: Drug: Ropivacaine
- Intervention (Experimental): Surgeon preforms inter-operative adductor canal block
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — For primary TKA, Ropivacaine is used in both arms, either performed intra-operatively by surgeon or post-operatively (ultrasound guided) by anesthesiologist.

SUMMARY:
The purpose of this study is to evaluate the efficacy of two methods of administering an adductor canal block (ACB) following total knee arthroplasty (TKA); intraoperative surgeon performed intra-articular adductor canal block (IACB) and anesthesiologist ultrasound guided ADC in the post-anesthesia recovery unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary TKA with underlying diagnosis of osteoarthritis
* ASA I - III
* Spinal anesthesia
* All patients will have cemented total knee utilizing a medial parapatellar approach with posterior stabilized or cruciate retaining implants. A tourniquet will be used in all cases.
* Patients must be between 18 and 80 years of age.
* Active and valid email address for the participant.

Exclusion Criteria:

* Allergy to anesthetics or study analgesic medications.
* Contraindication to regional anesthesia
* Non-english speaking
* ASA IV or greater
* Renal insufficiency with Cr > 2.0 or hepatic failure
* General or epidural anesthesia
* Sensory/motor disorder involving the operative limb
* Patients who consume preoperative opioids for pain control.
* Pregnant women
* Mentally disabled patients and patients with psychiatric disorders that would prevent them from properly understanding and evaluating an informed consent process.
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in visual analog scale pain score | Up to 6 weeks post-surgery
  The primary end point is the patients' reported visual analogue pain score (VAS). 0-100mm scale

SECONDARY OUTCOMES:
Change in range of motion | up to 6 weeks post-surgery
  Range of motion
Change in timed up and go | up to 6 weeks post-surgery
  Timed up and go
Change in daily opioid consumption | up to 6 weeks post-surgery
  daily opioid consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States